CLINICAL TRIAL: NCT02670369
Title: Investigating Sedentary Time in Aging: New Directions
Acronym: ISTAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5 K23 HL119352-1; 5K23HL119352 (NIH)
Record Dates: First submitted 2015-07-21; First posted 2016-02-01 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Sedentary Lifestyle
Keywords: Sedentary time; Sit-to-stand transitions
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sitting time prompt (Experimental): All participants will receive a prompting device (one-arm intervention).
  Interventions: Behavioral: Sitting time prompt

INTERVENTIONS:
Behavioral: Sitting time prompt — Participants will receive a device that prompts them to take breaks from sitting approximately every 15-20 minutes.

SUMMARY:
The investigators are doing a study to learn how to support patients aged 60+ in taking more breaks from sitting. The goal of the study is to find out if using commercially available devices are helpful in reducing sitting time.

DETAILED DESCRIPTION:
To date, no one has tested whether the prompting features of commercially available wrist-worn devices (e.g., Jawbone Up) improve breaks from sitting. Single case designs are a cost-effective way to conduct a controlled, randomized study that can inform larger intervention trials. Because the investigators are interested in ascertaining the effect of a very specific intervention on a very specific/single outcome, this study is well-suited to this approach.

The investigators will conduct iterative single case experimental studies using randomization tests. This design can help evaluate technologies for behavior change. To increase statistical power, the investigators opted to conduct an ABA study design (also termed a reversal design) where A is baseline and B is an intervention. Using randomization tests, the length of each A and B phase are determined to vary randomly in length prior to the beginning of each participant's experiment. The investigators will constrain the total time of each A and B phase to last a minimum of 5 days to provide adequate exposure to the A (measurement only) and B (intervention) conditions. The maximum total number of days participants will be enrolled is 28.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* BMI of 25+
* Ages 60+
* Continuously enrolled at Group Health for previous 12 months
* No record of death
* Not on the No Contact list
* Speaks, reads, and writes English
* Able to hold a conversation by phone (no hearing or other limitations)
* Self-reported ability to stand
* Self-reported ability to walk one block unassisted
* No history of an injury from a fall in past 3 months
* Work or retirement situations allows for taking breaks from sitting throughout the day
* Available for the study duration
* No unusual activities planned (e.g. travel, moving) during the study period
* Able to come to Group Health Capitol Hill/Central for measurement visits
* Willing to wear activity monitor (activPAL)
* Self-reports taking less than 4 breaks from sitting during an average hour
* Self-reports sitting more than 7 hours per day

Exclusion Criteria:

* Resides in long-term care, hospice care, or skilled nursing facility (previous 12 months)
* Wheelchair bound
* Diagnosis of dementia, serious mental health disorder, or substance use disorder (previous 24 months)
* Use of an assistive device

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Sit-to-stand transitions | up to 28 days
  Number of activPAL-measured sit-to-stand transitions measured at the day level

CONTACTS AND LOCATIONS:
Overall Officials: Dori E Rosenberg, PhD, MPH, Principal Investigator — Group Health Research Institute
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No